CLINICAL TRIAL: NCT02196220
Title: Ultrasonographic Assessment of Carpal Tunnel Syndrome in Children With Mucopolysaccharidosis and Comparison to Median Nerve Anatomy in Healthy Children.
Brief Title: Ultrasonographic Assessment of Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Hutchinson, M.D., University of Utah
Other Study IDs: 59910
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mucopolysaccharidosis are lysosomal storage disorders such as Hunter, Hurler, and Sanfilippo syndromes. These patients have a genetic enzyme deficiency that results in the inability to degrade glycosaminoglycans. The glycosaminoglycans accumulate in lysosomes causing cell enlargement and subsequent dysfunction. The accumulation occurs in all tissues including cartilage, joint capsule, and tendons and can lead to carpal tunnel syndrome, trigger digits, and various other orthopaedic manifestations [Van Heest, White]. These children often suffer from severe cognitive impairment and are often unable to communicate pain or numbness. Carpal tunnel syndrome is almost always present, but may not become apparent until symptoms are severe and loss of function has occurred. The current gold standard for diagnosis consists of electromyographic (EMG) and nerve conduction velocity (NCV) studies under sedation or general anesthetic [Khanna].

Primary Objective: The investigators plan to correlate EMG findings and median nerve cross-sectional area in children with mucopolysaccharidosis. The investigators hypothesis is that ultrasonography of the carpal tunnel in patients with mucopolysaccharidosis will prove to be an effective, reliable, and safe method to evaluate the median nerve, thus avoiding the need for EMG studies and anesthesia.

Secondary Objective: The investigators want to determine the cross-sectional area of the median nerve using ultrasonography in a cohort of healthy children, ages 3-12. The investigators plan to evaluate a cohort of healthy children to determine a normal cross-sectional area of the median nerve.

ELIGIBILITY:
Inclusion Criteria:

For the first arm of the study (25 participants):

* Children with mucopolysaccharidosis presenting to the senior author's clinic with signs or symptoms of carpal tunnel syndrome will be enrolled to receive both an EMG and carpal tunnel ultrasound of the upper extremities.

For the second arm of the study (100 participants):

* Healthy children ages 3-12 with no acute upper extremity trauma or history of mucopolysaccharidosis.
* 25 additional participants requested in case of inconclusive ultrasound results, patient removal, or other unusable results.

Exclusion Criteria:

First arm:

* Children with mucopolysaccharidosis who have undergone previous treatment for carpal tunnel syndrome.

Second arm:

* Acute (<3month) wrist or hand surgery/injuries.
* Unable to obtain parental consent or patient assent.
* History of mucopolysaccharidosis.
* Non-english speaking.
* Cognitive impairment.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study Size: *150 total which includes the following:
  Arm 1: 25 Children with mucopolysaccharidosis
  Arm 2: 100 Control Group - Healthy children ages 3-12 with no previous history of upper extremity trauma or history of mucopolysaccharidosis.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2013-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Median nerve cross-sectional area in children with mucopolysaccharidosis and a cohort of healthy children, ages 3-12. | 6-weeks after open carpal tunnel release

CONTACTS AND LOCATIONS:
Overall Officials: Douglas T Hutchinson, M.D., Principal Investigator — University of Utah Orthopedic Center; Amy Moeller, M.D., Principal Investigator — University of Utah Orthopedic Center
Locations (1):
- University of Utah/Primary Children's Medical Center, Salt Lake City, Utah, United States